CLINICAL TRIAL: NCT01755637
Title: A Single-dose, Two-centre, Randomized, Open-label, Two-way Crossover Bioequivalence Study of Two Kinds of AlbendazoleTablet Formulations in Healthy Chinese Adult Males
Brief Title: Bioequivalence Study of Albendazole 400 mg Tablets in Chinese Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: O7921353
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Results first posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-05

CONDITIONS: Helminthiasis
MeSH Terms: conditions — Helminthiasis | interventions — Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albendazole tablet (Aqua Based) (Experimental): Albendazole tablets 400 milligram (mg) manufactured under aqua based solvent condition taken orally with 200 millilitre (mL) of water as single dose treatment.
  Interventions: Drug: Albendazole
- Albendazole tablet (Alcohol Based) (Active Comparator): Albendazole tablets 400 mg manufactured under ethanol based solvent condition taken orally with 200 mL of water as single dose treatment.
  Interventions: Drug: Albendazole

INTERVENTIONS:
Drug: Albendazole — Albendazole tablets 400 mg

SUMMARY:
The purpose of the study is to compare the pharmacokinetic profiles of two Albendazole tablet formulations manufactured under the different granulation processes in healthy Chinese adult males.

DETAILED DESCRIPTION:
Due to the product manufacture process change in Albendazole oral formulation from ethanol based granulation process to aqua based granulation process, State Food and Drug Administration officially requested Tianjin Smith Kline and French Laboratories to carry out a Bioequivalence study to demonstrate bioequivalence between the manufacturing processes. This trial will be conducted to support the official requirement via the comparison of the pharmacokinetic profiles between both the drugs manufactured under the different processes.

After oral administration, Albendazole is quickly oxidized into its pharmacologically active metabolite, Albendazole sulphoxide (ABZ-SO. Due to extensive metabolism and limited absorption, plasma concentration of ABZ after oral administration was found to be too low to be measured. Thus, this trial will also compare the pharmacokinetic profiles of ABZ-SO manufactured using different solvents.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged from 18 years up to 40 years (inclusive).
2. Body mass index within the range of 19-24kg/m^2.
3. Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or physical examination.
4. Negative for serum hepatitis B surface antigen, hepatitis C antibody and antibody of HIV.

Exclusion Criteria:

1. Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
2. Substance abuse: Recent history (within the last year) of alcohol or other substance abuse or failed to pass drugs of abuse screen and/or alcohol screen test.
3. Disease

   1. Current or recurrent disease that could affect the action, absorption or distribution of the study medication or clinical or laboratory assessments (e.g. hepatic disorders, abnormal liver function tests, renal insufficiency, congestive heart failure);
   2. Current or relevant previous history of serious, severe or unstable physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the study medication or procedures;
   3. History of gastrointestinal bleeding or peptic ulcer;
   4. Asthma
   5. History of liver disease
4. Medication

   1. Use of any drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to dosing
   2. Current or regular use of any prescription or over-the-counter medication, any other ABZ containing products, and traditional Chinese medicine.
5. Smoking

   1. Subjects who are current smokers or non-smokers of less than 3 months;
   2. Prior (within seven days of dosing) or current use of any other nicotine containing products, including nicotine replacement therapy.
6. Blood

   1. Blood donation ≥ 500 ml within 90 days before the first study session.
   2. Plasma donation within the 90 days before the first study session.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-04; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- China (2):
  - Central Hospital of China Aerospace Corporation, Beijing, Beijing Municipality
  - Tongji Hospital, Medical College Huazhong, Wuhan, Hubei

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at two clinical sites in China.
Pre-assignment Details: Out of 123 screened participants, 54 did not meet the study criteria; 12 withdrew consent and one was lost to follow -up. Only 56 participants were randomized.
Groups:
- Albendazole (Aqua) First, Then Albendazole (Alcohol): Participants were orally administered with 400 milligram (mg) Albendazole tablets manufactured under aqua based solvent condition as single dose treatment, followed by single dose treatment of 400 mg albendazole tablets manufactured under ethanol based solvent conditions. A wash-out period of 7 days was maintained between treatment periods.
- Albendazole (Alcohol) First, Then Albendazole (Aqua): Participants were orally administered with 400 mg Albendazole tablets manufactured under ethanol based solvent condition as single dose treatment followed by 400 mg aqua based albendazole tablets. A wash-out period of 7 days was maintained between treatment periods.
Period: Period 1
Arm/Group | Albendazole (Aqua) First, Then Albendazole (Alcohol) | Albendazole (Alcohol) First, Then Albendazole (Aqua)
Started | 28 | 28
Completed | 28 | 27
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 2
Arm/Group | Albendazole (Aqua) First, Then Albendazole (Alcohol) | Albendazole (Alcohol) First, Then Albendazole (Aqua)
Started | 28 | 27
Completed | 28 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants were evaluated for baseline measures
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 56
Age Continuous [Mean (Standard Deviation); unit: Years] | 24.21 (2.715)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 56

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Time t [AUC(0-t)] of Albendazole.
Description: AUC (0-t) was evaluated using the trapezoid rule.
Time Frame: Blood samples were collected pre-dose 0 hour (hr) and post dose 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 7, 9, 12, 16, 24 and 36 hr
Population: The analysis was carried out per protocol population. Missing data was not imputed for evaluation.
Measure: Mean (Standard Deviation); unit: nanogram (ng).hr per milliliter (mL)
Groups:
- Experimental: Albendazole Tablet (Aqua Based): Participants were orally administered with 400 milligram (mg) Albendazole tablets manufactured under aqua based solvent condition as single dose treatment.
- Reference: Albendazole Tablet (Alcohol Based): Participants were orally administered with 400 mg Albendazole tablets manufactured under ethanol based solvent condition as single dose treatment.
Arm/Group | Experimental: Albendazole Tablet (Aqua Based) | Reference: Albendazole Tablet (Alcohol Based)
Number analyzed (Participants) | 55 | 55
nanogram (ng).hr per milliliter (mL) | 54.82 (51.56) | 48.07 (49.22)
Statistical Analysis 1: Comparison: Experimental: Albendazole Tablet (Aqua Based) vs Reference: Albendazole Tablet (Alcohol Based); The value was log-transformed and a linear mixed effects model was applied to this value, as the dependent variable, treatment, and period as fixed effects and participants as random effect; Test type: Non-Inferiority or Equivalence — The bioequivalence between the two products was concluded if the 90% CIs (based on log transformed data and anti-logged) for the ratio of the geometric means lie completely within the range 80%-125%; Geometric mean Ratio of treatments = 114.37, 90% CI 2-sided [100.49 to 130.16] — Geometric mean ratio of experimental and reference product was determined by exponentiating least-squares means of log-transformed value

2. Primary Outcome: AUC [0-infinity (Inf)] of Albendazole
Description: AUC (0-inf) was evaluated using the trapezoid rule.
Time Frame: Blood samples were collected pre-dose at 0 hr and post dose at 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 7, 9, 12, 16, 24 and 36 hr
Population: The analysis was carried out per protocol population. Missing data was not imputed for evaluation.
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Groups:
- Experimental: Albendazole Tablet (Aqua Based): Participants were orally administered with 400 mg Albendazole tablets manufactured under aqua based solvent condition as single dose treatment.
Arm/Group | Experimental: Albendazole Tablet (Aqua Based) | Reference: Albendazole Tablet (Alcohol Based)
Number analyzed (Participants) | 19 | 16
ng.hr/mL | 69.55 (80.44) | 67.19 (84.74)
Statistical Analysis 1: Comparison: Experimental: Albendazole Tablet (Aqua Based) vs Reference: Albendazole Tablet (Alcohol Based); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio of treatments = 107.41, 90% CI 2-sided [69.03 to 167.13] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Maximum Observed Plasma Concentration [Cmaximum (Max)] of Albendazole
Description: Cmax was depicted from plasma concentration of Albendazole.
Time Frame: as for outcome 2
Population: The analysis was carried out per protocol population. Missing data was not imputed for evaluation.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Experimental: Albendazole Tablet (Aqua Based) | Reference: Albendazole Tablet (Alcohol Based)
Number analyzed (Participants) | 55 | 56
ng/mL | 14.76 (15.88) | 14.58 (16.93)
Statistical Analysis 1: Comparison: Experimental: Albendazole Tablet (Aqua Based) vs Reference: Albendazole Tablet (Alcohol Based); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The bioequivalence between the two products was concluded if the 90% CIs (based on log transformed data and anti-logged) for the ratio of the geometric means lie completely within the range of 70% -143%; Geometric mean ratio of treatments = 111.28, 90% CI 2-sided [94.76 to 130.68] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Albendazole
Description: Tmax was time at which Cmax of Albendazole was reached.
Time Frame: as for outcome 2
Population: The analysis was carried out per protocol population. Participants were excluded where the baseline concentration was greater than 5% of Cmax.
Measure: Median (Full Range); unit: hr
Arm/Group | Experimental: Albendazole Tablet (Aqua Based) | Reference: Albendazole Tablet (Alcohol Based)
Number analyzed (Participants) | 55 | 56
hr | 1.50 [0.5 to 4.0] | 1.00 [0.5 to 3.0]
Statistical Analysis 1: Comparison: Experimental: Albendazole Tablet (Aqua Based) vs Reference: Albendazole Tablet (Alcohol Based); The null hypothesis considered that there is no median within-subject difference between two treatment groups; Test type: Superiority or Other; p = 0.0011, Wilcoxon signed rank test; The values were not adjusted for this non-parametric analysis; Median Difference (Final Values) = 0.0167 — The median difference was calculated as = (Experimental-Reference)

5. Secondary Outcome: AUC (0-t) of Active Metabolite - Albendazole Sulphoxide
Description: AUC (0-t) of Albendazole i.e. Albendazole sulphoxide was evaluated using the trapezoid rule.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Groups:
- Experimental: Albendazole Sulphoxide Tablet (Aqua Based): Participants were orally administered with 400 milligram (mg) Albendazole sulphoxide tablets manufactured under aqua based solvent condition as single dose treatment.
- Reference: Albendazole Sulphoxide Tablet (Alcohol Based): Participants were orally administered with 400 mg Albendazole sulphoxide tablets manufactured under ethanol based solvent condition as single dose treatment.
Arm/Group | Experimental: Albendazole Sulphoxide Tablet (Aqua Based) | Reference: Albendazole Sulphoxide Tablet (Alcohol Based)
Number analyzed (Participants) | 55 | 55
ng.hr/mL | 2563.90 (1108.19) | 2290.14 (944.72)
Statistical Analysis 1: Comparison: Experimental: Albendazole Sulphoxide Tablet (Aqua Based) vs Reference: Albendazole Sulphoxide Tablet (Alcohol Based); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio of treatments = 112.05, 90% CI 2-sided [103.65 to 121.12] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: AUC (0-inf) of Active Metabolite - Albendazole Sulphoxide
Description: AUC (0-inf) of Albendazole sulphoxide was evaluated using the trapezoid rule.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Groups:
- Experimental: Albendazole Sulphoxide Tablet (Aqua Based): Participants were orally administered with 400 mg Albendazole sulphoxide tablets manufactured under aqua based solvent condition as single dose treatment.
Arm/Group | Experimental: Albendazole Sulphoxide Tablet (Aqua Based) | Reference: Albendazole Sulphoxide Tablet (Alcohol Based)
Number analyzed (Participants) | 43 | 45
ng.hr/mL | 3263.88 (1456.41) | 2829.77 (1128.06)
Statistical Analysis 1: Comparison: Experimental: Albendazole Sulphoxide Tablet (Aqua Based) vs Reference: Albendazole Sulphoxide Tablet (Alcohol Based); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Geometric mean ratio of treatments = 113.10, 90% CI 2-sided [103.40 to 123.71] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Cmax of Active Metabolite - Albendazole Sulphoxide
Description: Cmax was depicted from plasma concentration of Albendazole.
Time Frame: as for outcome 2
Population: The analysis was carried out per protocol population. Missing data was not imputed for evaluation.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Experimental: Albendazole Sulphoxide Tablet (Aqua Based) | Reference: Albendazole Sulphoxide Tablet (Alcohol Based)
Number analyzed (Participants) | 55 | 56
ng/mL | 221.45 (105.87) | 199.99 (108.89)
Statistical Analysis 1: Comparison: Experimental: Albendazole Sulphoxide Tablet (Aqua Based) vs Reference: Albendazole Sulphoxide Tablet (Alcohol Based); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Geometric mean ratio of treatments = 114.33, 90% CI 2-sided [102.99 to 126.93] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the first dosage of the session one, and until 5 days following last administration of the investigational product.
Groups:
- Albendazole Tablet (Aqua Based): Participants were orally administered with 400 mg Albendazole tablets manufactured under aqua based solvent condition as single dose treatment.
- Albendazole Tablet (Alcohol Based): Participants were orally administered with 400 mg Albendazole tablets manufactured under ethanol based solvent condition as single dose treatment.
Arm/Group | Albendazole Tablet (Aqua Based) | Albendazole Tablet (Alcohol Based)
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 1/55 | 4/56
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albendazole Tablet (Aqua Based) (N=55) | Albendazole Tablet (Alcohol Based) (N=56)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Gamma-Glutamyl Transferase Increased (Investigations) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Albuminuria (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.